CLINICAL TRIAL: NCT02428842
Title: Biomarker Evaluation in Advanced Stage Cervical Cancer by an International Working Group. Tumor Stages (1B1 - 4)
Acronym: BIO-RAIDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IC 2013-02 BIO-RAIDs
Record Dates: First submitted 2015-02-10; First posted 2015-04-29 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; Tumor biopsies; Standard treatment; Molecular profile; Next Generation Sequencing
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tumor biopsies and blood sampling (Other): Patient will undergo standard care with tumor and blood sampling before and after treatment.
  Blood and tumor sampling will also be performed at disease progression/relapse.
  Interventions: Procedure: Tumor biopsies; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Tumor biopsies — Tumor biopsies will be performed before and after treatment.
Procedure: Blood sampling — Blood sampling will be performed before and after treatment.

SUMMARY:
Prospective Multicentric European trial for Cervical cancer, not previously treated, with tumour biopsies, and blood collection for molecular analysis at predetermined time points.

ELIGIBILITY:
Inclusion Criteria:

1. No prior treatment for cervical cancer.
2. FIGO Stage IB1 to IVB; all histological subtypes (excluding neuro-endocrine type).
3. Pelvic MRI available or planned before the start of treatment, , if FIGO ≥ IB2. and optional for IB1 stage
4. Possibility to communicate imaging data by CD-ROM (format DICOM 3.0 or more).
5. Disease amenable to biopsy (3 tumour samples are mandatory prior to treatment).
6. Age ≥ 18 years.
7. ECOG (Eastern Cooperative Oncology Group) 0-2.
8. Life expectancy > 6 months.
9. Patient eligible for standard treatment (according to standards of each center).
10. Patient having health care insurance.
11. Informed and signed consent by patient.

(DICOM = Digital Imaging and Communications in Medicine)

Exclusion Criteria:

1. Patient enrolled in a clinical trial involving an investigative new agent.
2. Co morbidity, preventing patient to tolerate the proposed standard treatment.
3. Past history of invasive cancer over the 5 years preceding entry in the present trial (except basal cell carcinoma and carcinoma in situ of the cervix).
4. Impossibility to carry out evaluation by MRI (patient claustrophobic, pacemaker, metallic implant, non availability, other), ), if FIGO ≥ IB2 .
5. Patient deprived from ability to decide on her own.
6. Patient unable to have a regular follow up for geographical, social or psychological reasons.
7. Pregnancy or patient old enough to procreate and not using effective contraceptive method.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2013-10-24 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Correlation between tumor biological profile and treatment response. | up to 6 months
  Dominant mutations and activation pathways in cervical cancers is assessed from tumor biopsies.

SECONDARY OUTCOMES:
Progression Free Survival evaluation | up to 18 months
  Number of patient with no local/metastasis relapse 18 months after end of primary treatment course.
Standard treatment description (Description of primary treatment course regarding : - Initial FIGO ( International Federation of Gynecology and Obstetrics ) staging at baseline - Geographic location(country) | up to six months
  Description of primary treatment course regarding :
  * Initial FIGO ( International Federation of Gynecology and Obstetrics
    ) staging at baseline
  * Geographic location(country)
Standard treatment's side effects description (assessed by compiling grade 3 and 4 sides effects during and after treatment (according to NCI CTCAE v4.03 scale - National Cancer Institute Common Toxicity Criteria for Adverse Effects) | up to 6 months
  Description of standard treatment's side effects will be assessed by compiling grade 3 and 4 sides effects during and after treatment (according to NCI CTCAE v4.03 scale
Molecular tumor alterations description (Description of molecular tumor alterations regarding geographic location (country) | up to 24 months
  Description of molecular tumor alterations regarding geographic location (country)

CONTACTS AND LOCATIONS:
Locations (24):
- France (17):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil - CHI Créteil, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Régional du Cancer de Montpellier - Val D'Aurelle, Montpellier
  - Institut de Cancérologie de Lorraine - ICL, Nancy
  - Institut de Cancérologie de l'Ouest - RENE GAUDUCHEAU, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Insitut Curie, Paris
  - Hôpital Tenon, Paris
  - Institut René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancérologie de Lorraine- ICL NANCY, Vandœuvre-lès-Nancy
  - Institut de Cancerologie Gustave Roussy, Villejuif
  - Groupe Hospitalier Bichat, Paris, Île-de-France Region
- Mhh Hanover - Hanover Medical School, Hanover, Germany
- Netherlands (2):
  - Amsterdam Medical Center (AMC), Amsterdam, Meibergdreef
  - Netherland Cancer Institute - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam
- Romania (3):
  - Teo Health S.A. - Spitalul Sf. Constantin, Brasov
  - Spitalul Clinic Municipal "Gavril Curteanu", Oradea
  - Clinica de radioterapie, Timișoara
- Clinic for operative oncology, Institute of oncology of Vojvodina, Kamenitz, Serbia

REFERENCES:
- [Derived] Chouchane-Mlik O, Oniga A, Latouche A, Halladjian M, Kleine-Borgmann FB, Gerardy JJ, Mittelbronn M, Kamal M, Scholl SM. Systematic assessment of tumor necrosis at baseline in cervical cancer - An independent factor associated with poor outcome. Hum Pathol. 2024 Jan;143:62-70. doi: 10.1016/j.humpath.2023.12.003. Epub 2023 Dec 20. PMID 38135059
- [Derived] Ngo C, Samuels S, Bagrintseva K, Slocker A, Hupe P, Kenter G, Popovic M, Samet N, Tresca P, von der Leyen H, Deutsch E, Rouzier R, Belin L, Kamal M, Scholl S; RAIDs consortium http://www.raids-fp7.eu/. From prospective biobanking to precision medicine: BIO-RAIDs - an EU study protocol in cervical cancer. BMC Cancer. 2015 Nov 4;15:842. doi: 10.1186/s12885-015-1801-0. PMID 26531748